CLINICAL TRIAL: NCT06870630
Title: Standard Versus Oesophago-gastric Junction Complex Myotomy for Treatment naïve Type 2 Achalasia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Director, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POEMUSM
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Diseases
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Per oral endoscopy myotomy for standard myotomy (Active Comparator): Standard myotomy is muscle fibers cutting in esophagus more than 7 cms
  Interventions: Device: Per oral endoscopy myotomy
- Per oral endoscopy myotomy for esophago gastric junction myotomy (Sham Comparator): Myotomy is muscle fibers cutting in esophagus less than 3 cms.
  Interventions: Device: Per oral endoscopy myotomy

INTERVENTIONS:
Device: Per oral endoscopy myotomy — Poem procedure is meant for cutting of circular and longitudinal muscle fibers in esophagus to reduce the symptoms of dysphagia, regurgitation and chestpain, weight loss.

SUMMARY:
- Consecutive eligible patients will be randomized in a 1:1 ratio to esophagogastric complex only myotomy or standard myotomy groups. Randomization is done according to the computer-generated algorithm. A clinical research coordinator will prepare the sealed randomization envelops and will hand over to the operating endoscopists before the beginning of the procedure. Written informed consent will be obtained from all participants. In this study, the participants and the care-provider assessing the clinical response to the POEM procedure at 3months will be blinded to the allocation.

DETAILED DESCRIPTION:
. Primary objective -

• To study the incidence of true reflux on 24 hour pH analysis with manual study.

Secondary objective -

* To analyse treatment success which is defined as Eckdart score < 3 at follow up assessment ( 3rd month)
* To analyse the recovery of peristalsis after POEM using High resolution manometry
* To study total procedure time , intra operative adverse effects and duration of hospital stay.
* Severity of oesophagitis
* Presence of GERD symptoms based on GERD questionnaire & Quality of life questionaire post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years
* Diagnosis of Type 2 Achalasia cardia based on High resolution manometry.

Exclusion Criteria:

* Patients with Type 1 & 3 ACHALASIA CARDIA
* Patients with previous endoscopic or surgical treatment for achalasia
* Patients with standard exclusion criteria for POEM procedure such as contraindication to general anesthesia, coagulopathy (international normalized ratio > 1.5, platelet count < 50 000/μL), portal hypertension, pregnancy, breast feeding women, and diffuse scarring in the esophagus due to previous surgery or radiation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of true reflux based on 24-hour pH impedence | 3 months
  Reflux parameters in percent are noted in impedence report like acidic and non acidic refluxes
Integrated Relaxation Pressure (IRP) at High resolution manometry test | 3 months
  IRP in mm Hg measures pressure in the esophagus

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Dr Ramchandani, MBBS MD, Study Director — AIG Hospitals; Zaheer Dr Nabi, MBBS MD, Principal Investigator — AIG Hospitals; Pradev Dr Inovolu, MBBS MD, Principal Investigator — AIG Hospitals
Locations (1):
- Asian Institute of Gastroenterology /Aig Hospitals, Hyderabad, Telangana, India